CLINICAL TRIAL: NCT06890286
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 2-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between Single Oral Administration of BR3006 and Co-administration of BR3006A, BR3006B and BR3006C in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between Single Oral Administration of BR3006 and Co-administration of BR3006A, BR3006B and BR3006C in Healthy Adult Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPMC-CT-102
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR3006 (Experimental)
  Interventions: Drug: BR3006
- BR3006A+BR3006B+BR3006C (Active Comparator)
  Interventions: Drug: BR3006A; Drug: BR3006B; Drug: BR3006C

INTERVENTIONS:
Drug: BR3006 — One tablet administered alone
  Arms: BR3006
Drug: BR3006A — One tablet administered alone
  Arms: BR3006A+BR3006B+BR3006C
Drug: BR3006B — One tablet administered alone
  Arms: BR3006A+BR3006B+BR3006C
Drug: BR3006C — One tablet administered alone
  Arms: BR3006A+BR3006B+BR3006C

SUMMARY:
The purpose of this clinical study is to evaluate the pharmacokinetics and safety between single oral administration of BR3006 and co-administration of BR3006A, BR3006B and BR3006C in healthy adult volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Those who have body mass index (BMI) of 18.0kg/m2 to 30.0kg/m2 at screening visit.

  * For men, Those who weigh 55 kg or more
  * For women, Those who weigh 50 kg or more
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial* from the date of consent to 14 days after the last administration and disagree to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of non hormonal intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken ethical drugs, over the counter drugs, herbal medicines, health functional foods concerned about affecting this clinical trial within 10 days before the first administration date. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have a medical history of gastrointestinal resection (Except for simple appendectomy, hernia surgery) or gastrointestinal diseases that may affect the absorption of drugs.
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months before the first administration date(However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* In the case of a female subject, pregnant woman or those suspected pregnancy or lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-96 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time t
Cmax | 0-96 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No